CLINICAL TRIAL: NCT04096586
Title: Effects of Watermelon Consumption on Satiety and Digestive Health
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: San Diego State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: HS-2019-0103
Record Dates: First submitted 2019-09-18; First posted 2019-09-20 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Satiety

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Red juice (Active Comparator): Subjects consume 8 fl oz of red juice daily for 8 weeks
  Interventions: Other: Red juice
- Watermelon juice (Experimental): Subjects consume 8 fl oz of watermelon juice daily for 8 weeks
  Interventions: Other: Watermelon juice

INTERVENTIONS:
Other: Red juice — To determine the effects of red juice on satiety and gut health
  Arms: Red juice
Other: Watermelon juice — To determine the effects of watermelon juice on satiety and gut health
  Arms: Watermelon juice

SUMMARY:
The objective of the proposed research is to determine the effects of watermelon (fruit and rind blenderized) on satiety, metabolic markers, bowel habits, microbiome and weight management in children and adults

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy subjects

Exclusion Criteria:

* Smoker
* Pregnant woman
* Required dietary supplement use
* Required medication of metabolic disorders
* Allergy to watermelon

Ages: 10 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 80 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change of satiety | 0 and 20, 40, 60, 90 and 120 minutes post juice consumption
  Change of hunger feeling (appetite) will be examined using visual analog scale (0-10), 0 least and 10 greatest
Change of glucose level | 0 and 20, 40, 60, 90 and 120 minutes post juice consumption
  Change of blood glucose level will be determined to examine effects of watermelon juice consumption vs red juice
Change of insulin level | 0 and 20, 40, 60, 90 and 120 minutes post juice consumption
  Change of blood insulin level will be determined to examine effects of watermelon juice consumption vs red juice
Change of triglyceride level | Baseline and week 8
  Change of triglyceride level with watermelon juice consumption vs red juice consumption

SECONDARY OUTCOMES:
Change of alpha diversity in microbiome | Baseline and week 8
  Change of alpha diversity in micriobiome with watermelon juice consumption vs red juice consumption

CONTACTS AND LOCATIONS:
Locations (1):
- School of Exercise and Nutritional Sciences, SDSU, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No